CLINICAL TRIAL: NCT02568345
Title: Sugammadex ED90 Dose to Reverse the Rocuronium Blockade in the Obese Patients
Brief Title: Sugammadex ED90 Dose in the Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Mauro Prado da Silva, MD, Staff, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191.837
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Incomplete Reversal of Neuromuscular Block
Keywords: Dose-Response Relationship; Drug; Obesity; Cyclodextrins
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sugammadex ED90 (Experimental): Sequential design method up-and-down of the biased coin aimed to determine the minimum effective dose in 90% of patients (ED90).
  The following doses were chosen: 2.0 mg/kg, 2.2 mg/kg, 2.4 mg/kg, 2.6 mg/kg, 2.8 mg/kg.
  Interventions: Drug: sugammadex ED90

INTERVENTIONS:
Drug: sugammadex ED90 — The first patient received the dose of 2.4 mg/kg and if there was a negative response, the next patient would be allocated to receive the next higher dose of 2.6 mg/kg.
  In case that 2.4 mg/kg did produce a positive response, the next patient would be randomized with 10% of probability to receive the next dose of 2.2 mg/kg or 90% probability to receive the same dose of 2.4 mg/kg.
  Other Names: ED90

SUMMARY:
The purpose of this study is to determine the minimum effective dose of sugammadex, an antagonist of neuromuscular blockade used during anesthesia practice, in obese patients, considering that sugammadex is indicated in adults with normal weight at a dose of 2 mg/kg but no studies were found with obese patients.

DETAILED DESCRIPTION:
Prospective study with the sequential design method up-and-down of the biased coin aimed to determine the minimum effective dose in 90% of patients (ED90).

The following doses were chosen: 2.0 mg.kg-1, 2.2 mg.kg-1, 2.4 mg.kg-1, 2.6 mg.kg-1, 2.8 mg.kg-1.

The complete reversal of moderate rocuronium-induced neuromuscular blockade (NMB) considered a T4/T1 ratio ≥ 0.9 with the peripheral nerve stimulator and accelerometer (monitor of sequential electric stimuli) "train-of-four" (TOF).

After induction of general anesthesia and the calibration of the peripheral nerve stimulator and accelerometer, rocuronium 0.6 mg.kg-1 was injected.

Continuous intravenous infusion of the anesthetics propofol and remifentanil, and intermittent bolus of rocuronium were offered throughout the procedure.

ELIGIBILITY:
Inclusion Criteria:

* a body mass index ≥ 40 kg/m2
* bariatric surgery
* informed consent signed

Exclusion Criteria:

* history of neuromuscular diseases,
* use of drugs that could interfere with neuromuscular transmission,
* allergy to neuromuscular agents of the aminosteroids class,
* anticipated difficulty in airway management,
* renal failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lígia Andrade ST Mathias, MD, Ph.D, Study Director — Full professor

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] 1983 metropolitan height and weight tables. Stat Bull Metrop Life Found. 1983 Jan-Jun;64(1):3-9. No abstract available. PMID 6623350
- [Background] Abernethy DR, Greenblatt DJ, Divoll M, Smith RB, Shader RI. The influence of obesity on the pharmacokinetics of oral alprazolam and triazolam. Clin Pharmacokinet. 1984 Mar-Apr;9(2):177-83. doi: 10.2165/00003088-198409020-00005. PMID 6143633
- [Background] Blouin RA, Kolpek JH, Mann HJ. Influence of obesity on drug disposition. Clin Pharm. 1987 Sep;6(9):706-14. PMID 3315402
- [Background] de Boer HD, Driessen JJ, Marcus MA, Kerkkamp H, Heeringa M, Klimek M. Reversal of rocuronium-induced (1.2 mg/kg) profound neuromuscular block by sugammadex: a multicenter, dose-finding and safety study. Anesthesiology. 2007 Aug;107(2):239-44. doi: 10.1097/01.anes.0000270722.95764.37. PMID 17667567
- [Background] Donati F. Sugammadex: a cyclodextrin to reverse neuromuscular blockade in anaesthesia. Expert Opin Pharmacother. 2008 Jun;9(8):1375-86. doi: 10.1517/14656566.9.8.1375. PMID 18473711
- [Background] Duffull SB, Dooley MJ, Green B, Poole SG, Kirkpatrick CM. A standard weight descriptor for dose adjustment in the obese patient. Clin Pharmacokinet. 2004;43(15):1167-78. doi: 10.2165/00003088-200443150-00007. PMID 15568893
- [Background] Epemolu O, Bom A, Hope F, Mason R. Reversal of neuromuscular blockade and simultaneous increase in plasma rocuronium concentration after the intravenous infusion of the novel reversal agent Org 25969. Anesthesiology. 2003 Sep;99(3):632-7; discussion 6A. doi: 10.1097/00000542-200309000-00018. PMID 12960547
- [Background] Janmahasatian S, Duffull SB, Ash S, Ward LC, Byrne NM, Green B. Quantification of lean bodyweight. Clin Pharmacokinet. 2005;44(10):1051-65. doi: 10.2165/00003088-200544100-00004. PMID 16176118
- [Background] Mosteller RD. Simplified calculation of body-surface area. N Engl J Med. 1987 Oct 22;317(17):1098. doi: 10.1056/NEJM198710223171717. No abstract available. PMID 3657876
- [Background] Nicholson WT, Sprung J, Jankowski CJ. Sugammadex: a novel agent for the reversal of neuromuscular blockade. Pharmacotherapy. 2007 Aug;27(8):1181-8. doi: 10.1592/phco.27.8.1181. PMID 17655516
- [Background] Pai MP, Paloucek FP. The origin of the "ideal" body weight equations. Ann Pharmacother. 2000 Sep;34(9):1066-9. doi: 10.1345/aph.19381. PMID 10981254
- [Background] Renes SH, van Geffen GJ, Rettig HC, Gielen MJ, Scheffer GJ. Minimum effective volume of local anesthetic for shoulder analgesia by ultrasound-guided block at root C7 with assessment of pulmonary function. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):529-34. doi: 10.1097/AAP.0b013e3181fa1190. PMID 20975468
- [Background] Sorgenfrei IF, Norrild K, Larsen PB, Stensballe J, Ostergaard D, Prins ME, Viby-Mogensen J. Reversal of rocuronium-induced neuromuscular block by the selective relaxant binding agent sugammadex: a dose-finding and safety study. Anesthesiology. 2006 Apr;104(4):667-74. doi: 10.1097/00000542-200604000-00009. PMID 16571960
- [Background] Stylianou M, Flournoy N. Dose finding using the biased coin up-and-down design and isotonic regression. Biometrics. 2002 Mar;58(1):171-7. doi: 10.1111/j.0006-341x.2002.00171.x. PMID 11890313
- [Result] Demirkaya M, Kelsaka E, Sarihasan B, Bek Y, Ustun E. The optimal dose of remifentanil for acceptable intubating conditions during propofol induction without neuromuscular blockade. J Clin Anesth. 2012 Aug;24(5):392-7. doi: 10.1016/j.jclinane.2011.11.006. PMID 22748212
- [Result] Garrett-Mayer E. The continual reassessment method for dose-finding studies: a tutorial. Clin Trials. 2006;3(1):57-71. doi: 10.1191/1740774506cn134oa. PMID 16539090
- [Result] George RB, McKeen D, Chaplin AC, McLeod L. Up-down determination of the ED(90) of oxytocin infusions for the prevention of postpartum uterine atony in parturients undergoing Cesarean delivery. Can J Anaesth. 2010 Jun;57(6):578-82. doi: 10.1007/s12630-010-9297-1. Epub 2010 Mar 18. PMID 20238255
- [Result] Gupta PK, Hopkins PM. Effect of concentration of local anaesthetic solution on the ED(5)(0) of bupivacaine for supraclavicular brachial plexus block. Br J Anaesth. 2013 Aug;111(2):293-6. doi: 10.1093/bja/aet033. Epub 2013 Mar 26. PMID 23533252
- [Result] Hammer GB, Litalien C, Wellis V, Drover DR. Determination of the median effective concentration (EC50) of propofol during oesophagogastroduodenoscopy in children. Paediatr Anaesth. 2001;11(5):549-53. doi: 10.1046/j.1460-9592.2001.00731.x. PMID 11696118
- [Result] Hennebry MC, Stocks GM, Belavadi P, Barnes J, Wray S, Columb MO, Lyons G. Effect of i.v. phenylephrine or ephedrine on the ED50 of intrathecal bupivacaine with fentanyl for caesarean section. Br J Anaesth. 2009 Jun;102(6):806-11. doi: 10.1093/bja/aep095. Epub 2009 May 2. PMID 19411667
- [Result] Kodaka M, Suzuki T, Maeyama A, Koyama K, Miyao H. Gender differences between predicted and measured propofol C(P50) for loss of consciousness. J Clin Anesth. 2006 Nov;18(7):486-9. doi: 10.1016/j.jclinane.2006.08.004. PMID 17126774
- [Result] Llaurado S, Sabate A, Ferreres E, Camprubi I, Cabrera A. Sugammadex ideal body weight dose adjusted by level of neuromuscular blockade in laparoscopic bariatric surgery. Anesthesiology. 2012 Jul;117(1):93-8. doi: 10.1097/ALN.0b013e3182580409. PMID 22549697
- [Result] Pace NL, Stylianou MP. Advances in and limitations of up-and-down methodology: a precis of clinical use, study design, and dose estimation in anesthesia research. Anesthesiology. 2007 Jul;107(1):144-52. doi: 10.1097/01.anes.0000267514.42592.2a. PMID 17585226
- [Result] Stylianou M, Proschan M, Flournoy N. Estimating the probability of toxicity at the target dose following an up-and-down design. Stat Med. 2003 Feb 28;22(4):535-43. doi: 10.1002/sim.1351. PMID 12590412
- [Result] Taha AM, Abd-Elmaksoud AM. Lidocaine use in ultrasound-guided femoral nerve block: what is the minimum effective anaesthetic concentration (MEAC90)? Br J Anaesth. 2013 Jun;110(6):1040-4. doi: 10.1093/bja/aes595. Epub 2013 Feb 5. PMID 23384731
- [Result] Van Lancker P, Dillemans B, Bogaert T, Mulier JP, De Kock M, Haspeslagh M. Ideal versus corrected body weight for dosage of sugammadex in morbidly obese patients. Anaesthesia. 2011 Aug;66(8):721-5. doi: 10.1111/j.1365-2044.2011.06782.x. Epub 2011 Jun 21. PMID 21692760

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex ED90: Sequential design method up-and-down of the biased coin aimed to determine the minimum effective dose in 90% of patients (ED90).
  The following doses were chosen: 2.0 mg/kg, 2.2 mg/kg, 2.4 mg/kg, 2.6 mg/kg, 2.8 mg/kg.
  sugammadex ED90: The first patient received the dose of 2.4 mg/kg and if there was a negative response, the next patient would be allocated to receive the next higher dose of 2.6 mg/kg.
  In case that 2.4 mg/kg did produce a positive response, the next patient would be randomized with 10% of probability to receive the next dose of 2.2 mg/kg or 90% probability to receive the same dose of 2.4 mg/kg.
Period: Overall Study
Arm/Group | Sugammadex ED90
Started | 31
Treated at 2.2 mg/kg | 3 (patients: 6th, 20th, 26th)
Treated at 2.4 mg/kg | 25 (Patients: 1st-5th; 7th; 11th-15th; 21st-25th; 27th-31st)
Treated at 2.6 mg/kg | 3 (Patients: 8th-10th)
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sugammadex ED90
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [35 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 7
Region of Enrollment [Number; unit: participants]
  Brazil | 31
body mass index: kg.m^2 [Median (Inter-Quartile Range); unit: kg/m^2] | 49.3 [44.3 to 52.0]

OUTCOME MEASURES:

1. Primary Outcome: Sugammadex ED90
Description: Complete reversal of neuromuscular blockade occured when the patient had a TOF T4/T1 ≥ 0.9 within eight minutes of sugammadex infusion.
  The sequencial design method of up-and-down was applied to determine the minimum effective dose in 90% of patients (ED90). An effective dose is one that achieves complete reversal of neuromuscular blockade that is defined as a measure of TOF equal or higher than 0.9, or a relationship between T4 an T1 measure ≥ 0.9, within eight minutes of sugammadex infusion.
Time Frame: 8 minutes
Measure: Number (99% Confidence Interval); unit: mg/kg
Arm/Group | Sugammadex ED90
Number analyzed (Participants) | 31
mg/kg | 2.40 [2.20 to 2.60]
Statistical Analysis 1: Comparison: Sugammadex ED90; Test type: Superiority or Other; The isotonic regression functions through PAVA algorithm were used (pooled adjacent violators algorithm), to determine the ED90, and bootstrapping to calculate the respective 95% confidence interval with the statistical program R; isotonic regression functions through PA = 2.20

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Sugammadex ED90
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No